CLINICAL TRIAL: NCT04219488
Title: Comparison of the Effects of Neuromobilization and Conservative Rehabilitation Therapy on Pain, Grip Strength and Functional Status in Lateral Epicondylitis
Brief Title: Investigating the Effects of Neuromobilization in Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KaratayUK
Record Dates: First submitted 2019-12-31; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
Keywords: eccentric exercise; radial nerve mobilization
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromobilization group (Experimental): The neuromobilization group received a supervised home program plus radial nerve mobilization. Radial nerve mobilization exercises were performed by the physiotherapist for 3 days a week for 3 weeks. The patients in the neuromobilization group also performed self-neuromobilization exercises at home for 6 weeks. Supervised home program including patient education and eccentric exercises was administered three times daily for 6 weeks.
  Interventions: Other: Radial nerve mobilization; Other: Supervised home program
- Control group (Active Comparator): The control group received a supervised home program. Supervised home program including patient education and eccentric exercises was administered 3 times a day for 6 weeks.
  Interventions: Other: Supervised home program

INTERVENTIONS:
Other: Radial nerve mobilization
  Arms: Neuromobilization group
Other: Supervised home program

SUMMARY:
This study aimed to determine the effects of neuromobilization techniques and conservative rehabilitation therapy on pain, grip strength, and functional status in patients with lateral epicondylitis (LE). A total of 40 patients (26 females and 14 males; age: 42.80 ± 8.91 years) with a history of LE participated in the study. The patients were randomly assigned to two groups: the neuromobilization group and the control group. The neuromobilization group completed a 6-week conservative rehabilitation and radial nerve mobilization program, whereas the control group received conservative rehabilitation therapy only. Both groups underwent a 7-day weekly conservative home rehabilitation program. Pain severity, grip strength, pinch strength, joint mobility, and upper extremity functional level were assessed before treatment, at the third week, after treatment, and at the sixth week after treatment.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is a painful situation, which usually occurs due to the overuse of the wrist extensor muscles. The prevalence of LE is 1%-3% in both men and women, and it is highest in individuals aged >40 years. Pain and tenderness over the lateral epicondyle of the humerus at the origin of the common extensor tendon are the main characteristics. Different conservative treatment methods have been used for treating LE; however, no standard protocol has been documented in the literature. Physiotherapy programs have focused on relieving pain, controlling inflammation, and increasing muscle strength and endurance. The use of eccentric strengthening programs has been supported by current research. Eccentric exercises have been demonstrated to reduce pain and increase function in patients with LE. Recently, neuromobilization techniques have been employed in treating musculoskeletal problems and various compression syndromes. These techniques aimed to provide nerve gliding via joint movements wherein a therapist extends the nerve length in one joint while shortening the same in the adjacent joint. This tensioning technique increases the distance between each end of the nerve, and this neural elongation ability significantly decreases in patients with LE. Neuromobilization techniques have been also proposed to modulate central sensitization and peripheral pain mechanisms in musculoskeletal disorders. Given that central sensitization plays an important role in the increased nociceptive reflex and hyperalgesia in LE, inducing hypoalgesia via neuromobilization techniques may provide pain relief in the long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years
* A symptom duration of >3 months

Exclusion Criteria:

* Bilateral symptoms
* Rheumatologic diseases affecting the elbow and the wrist
* Musculoskeletal disorders due to connective tissue diseases
* Diffuse pain syndrome
* Cervical radiculopathy
* Nerve compression syndromes involving upper extremity
* Undergone surgery at the affected arm
* Received an LE treatment in the last 6 months
* An inability to perform the exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2014-12-15 (Actual); Study Completion 2015-01-05 (Actual)

PRIMARY OUTCOMES:
Pain severity | at the beginning of treatment
  Pain severity was measured using a 10-cm visual analog scale, labeled from 0 (no pain) to 10 (the worst pain), at rest, at night, and during daily activities
Pain severity | 3 weeks later
  Pain severity was measured using a 10-cm visual analog scale, labeled from 0 (no pain) to 10 (the worst pain), at rest, at night, and during daily activities
Pain severity | 6 weeks later
  Pain severity was measured using a 10-cm visual analog scale, labeled from 0 (no pain) to 10 (the worst pain), at rest, at night, and during daily activities
Pain severity | 12 weeks later
  Pain severity was measured using a 10-cm visual analog scale, labeled from 0 (no pain) to 10 (the worst pain), at rest, at night, and during daily activities
Grip strength | at the beginning of treatment
  Grip strength was measured using two different test methods: pain-free grip strength and maximum grip strength. Both tests were performed in the sitting position with the elbow flexed at 90° and in the standing position with the elbow extended at 0°. Both tests were performed using a calibrated hydraulic hand dynamometer® (Jamar, Bolingbrook IL).The measurements of both extremities were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kilograms (kg).
Grip strength | 3 weeks later
  Grip strength was measured using two different test methods: pain-free grip strength and maximum grip strength. Both tests were performed in the sitting position with the elbow flexed at 90° and in the standing position with the elbow extended at 0°. Both tests were performed using a calibrated hydraulic hand dynamometer® (Jamar, Bolingbrook IL).The measurements of both extremities were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kilograms (kg).
Grip strength | 6 weeks later
  Grip strength was measured using two different test methods: pain-free grip strength and maximum grip strength. Both tests were performed in the sitting position with the elbow flexed at 90° and in the standing position with the elbow extended at 0°. Both tests were performed using a calibrated hydraulic hand dynamometer® (Jamar, Bolingbrook IL).The measurements of both extremities were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kilograms (kg).
Grip strength | 12 weeks later
  Grip strength was measured using two different test methods: pain-free grip strength and maximum grip strength. Both tests were performed in the sitting position with the elbow flexed at 90° and in the standing position with the elbow extended at 0°. Both tests were performed using a calibrated hydraulic hand dynamometer® (Jamar, Bolingbrook IL).The measurements of both extremities were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kilograms (kg).
Tip pinch and key pinch | at the beginning of treatment
  Tip pinch and key pinch were measured using the "Baseline Mechanical Pinch Gauge" (FEI, White Plains, NY). Measurements were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kg.
Tip pinch and key pinch | 3 weeks later
  Tip pinch and key pinch were measured using the "Baseline Mechanical Pinch Gauge" (FEI, White Plains, NY). Measurements were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kg.
Tip pinch and key pinch | 6 weeks later
  Tip pinch and key pinch were measured using the "Baseline Mechanical Pinch Gauge" (FEI, White Plains, NY). Measurements were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kg.
Tip pinch and key pinch | 12 weeks later
  Tip pinch and key pinch were measured using the "Baseline Mechanical Pinch Gauge" (FEI, White Plains, NY). Measurements were repeated 3 times with a resting interval of 30 s between each measurement. The average of the three trials was recorded in kg.

SECONDARY OUTCOMES:
Wrist active range of motion (ROM)'s | at the beginning of treatment
  Wrist active ROMs, including flexion, extension, and radial and ulnar deviation were recorded in degrees by using a universal goniometer for each group.
Wrist active range of motion (ROM)'s | 3 weeks later
  Wrist active ROMs, including flexion, extension, and radial and ulnar deviation were recorded in degrees by using a universal goniometer for each group.
Wrist active range of motion (ROM)'s | 6 weeks later
  Wrist active ROMs, including flexion, extension, and radial and ulnar deviation were recorded in degrees by using a universal goniometer for each group.
Wrist active range of motion (ROM)'s | 12 weeks later
  Wrist active ROMs, including flexion, extension, and radial and ulnar deviation were recorded in degrees by using a universal goniometer for each group.
The functional status of the upper extremity | at the beginning of treatment
  The functional status of the upper extremity was evaluated using the Turkish version of the disabilities of the arm, shoulder and hand (DASH) questionnaire. The DASH questionnaire includes 30 items related to symptoms and activities of daily living. The total score is 100, and a higher score indicates a higher degree of disability.
The functional status of the upper extremity | 3 weeks later
  The functional status of the upper extremity was evaluated using the Turkish version of the disabilities of the arm, shoulder and hand (DASH) questionnaire. The DASH questionnaire includes 30 items related to symptoms and activities of daily living. The total score is 100, and a higher score indicates a higher degree of disability.
The functional status of the upper extremity | 6 weeks later
  The functional status of the upper extremity was evaluated using the Turkish version of the disabilities of the arm, shoulder and hand (DASH) questionnaire. The DASH questionnaire includes 30 items related to symptoms and activities of daily living. The total score is 100, and a higher score indicates a higher degree of disability.
The functional status of the upper extremity | 12 weeks later
  The functional status of the upper extremity was evaluated using the Turkish version of the disabilities of the arm, shoulder and hand (DASH) questionnaire. The DASH questionnaire includes 30 items related to symptoms and activities of daily living. The total score is 100, and a higher score indicates a higher degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Yılmaz, 1, Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)